CLINICAL TRIAL: NCT04133324
Title: Diagnosis Accuracy of the C-protein Reactive for the Detection of Anastomotic Leakage After Surgery for Digestive Cancer
Brief Title: C-protein Reactive for the Detection of Anastomotic Leakage After Surgery for Digestive Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moroccan Society of Surgery (Other)
Responsible Party: Principal Investigator, Anass Majbar, Study investigator, Moroccan Society of Surgery
Other Study IDs: CRP_study
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: C-Reactive Protein; Anastomotic Leak; Digestive System Neoplasm
MeSH Terms: conditions — Anastomotic Leak; Digestive System Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main group: One groupe in the study
  Interventions: Diagnostic Test: C-reactive protein

INTERVENTIONS:
Diagnostic Test: C-reactive protein — C-reactive protein at postoperative days four and two.

SUMMARY:
The aim of this study is to investigate the diagnostic accuracy of the C Protein Reactive (CRP) for the detection of Anastomotic leakage after surgery for digestive cancer. The standard protocol in our unit is to measure the CRP on the second and fourth postoperative day.

The main aim of the study is to investigate the diagnostic accuracy of the ratio CRP on the fourth postoperative day on CRP on the second postoperative day (CRP_D4/CRP_D2). Secondary outcomes are the diagnosis accuracy of the CRP_D4 and CRP_D2.

DETAILED DESCRIPTION:
The occurrence of anastomotic fistula (AF) is the most feared complication after digestive cancer surgery. It is responsible for high morbidity and accounts for more than a third of the deaths observed. The rate of anastomotic fistula reported in the literature varies between 1 and 40% according to the definition chosen by the authors. In the literature, the occurrence of the anastomotic fistula is responsible for a mortality rate of 4% and an overall morbidity of 35%. In the short term, the anastomotic fistula can put the patient's vital prognosis at risk by its septic consequences. Also, it is responsible for increasing the length of stay and costs. In the longer term, anastomotic fistula affects the functional prognosis of the patient as well as oncology in patients operated for cancer.

Early rehabilitation becomes a standard in colorectal surgery, with exits around the 5th postoperative day. Anastomotic fistulas and their complications may appear well beyond. The diagnosis is made on average around 6-7 postoperative days. At an early stage, clinical signs are inconsistent and not very specific. Anastomotic fistula can manifest itself in a variety of clinical presentations, ranging from no symptoms to life-threatening septic shock. Routine imaging is neither reliable nor cost-effective for the detection of anastomotic fistulas and has the disadvantage of radiation.

It is necessary to find an intraperitoneal infection marker with a high negative predictive value. This is particularly important in the era of early rehabilitation, allowing for safe patient discharge with a low risk of readmission. C-reactive protein (CRP) has already shown its utility in the early detection of infections after digestive surgery, however, because of conflicting results, no clear recommendations are established in the literature.

Our study aims are to investigate the diagnostic accuracy of the postoperative CRP trajectory as an approach to eliminate the diagnosis of anastomotic fistula and to try to establish an optimal threshold with high sensitivity and negative predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Surgical resection for digestive cancer
* Creation of anastomosis.
* at least one measurement of CRP at the second and/or fourth postoperative day.

Exclusion Criteria:

* Surgical resection without anastomosis creation
* No measurement of CRP on the second or the fourth postoperative day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who will undergo surgical resection for digestive cancer with the creation of anastomosis will be included. The standard protocol in our unit is to measure the CRP at the second and fourth postoperative days for early detection of anastomotic leakage.
  The following information will be recorded: age, gender, type of surgery, type of anastomosis, postoperative morbidity according to Clavien Grade, anastomotic leakage occurrence, infectious complications.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
CRP_D4/CRP_D2 | 30 days after surgery
  Diagnosis accuracy of the ratio CRP at the fourth on the second postoperative day after surgical resection for digestive cancer, using the receiving operating curve, sensibility, specificity, positive predictive value, and negative predictive value.
CRP_D4/CRP_D2 Colorectal | 30 days after surgery
  Diagnosis accuracy of the ratio CRP at the fourth on the second postoperative day after surgical resection for colorectal cancer, using the receiving operating curve, sensibility, specificity, positive predictive value, and negative predictive value.

SECONDARY OUTCOMES:
CRP_D4 | 30 days after surgery
  Diagnosis accuracy of the ratio CRP at the fourth postoperative day after surgical resection for digestive cancer, using the receiving operating curve, sensibility, specificity, positive predictive value, and negative predictive value.
CRP_D4 colorectal | 30 days after surgery
  Diagnosis accuracy of the ratio CRP at the fourth postoperative day after surgical resection for colorectal cancer, using the receiving operating curve, sensibility, specificity, positive predictive value, and negative predictive value.
CRP_D2 | 30 days after surgery
  Diagnosis accuracy of the ratio CRP at the second postoperative day after surgical resection for digestive cancer, using the receiving operating curve, sensibility, specificity, positive predictive value, and negative predictive value.
CRP_D2 colorectal | 30 days after surgery
  Diagnosis accuracy of the ratio CRP at the second postoperative day after surgical resection for colorectal cancer, using the receiving operating curve, sensibility, specificity, positive predictive value, and negative predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Anass Majbar, MD, Principal Investigator — National Institute of Oncology
Locations (1):
- National Institute of Oncology, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: Undecided